CLINICAL TRIAL: NCT01999517
Title: Contrast Nephropathy and Nitrates
Acronym: CoNaN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: Florida Heart Research Institute (Other)
Responsible Party: Principal Investigator, Gervasio Lamas, MD, Chied of Medicine, Chair of Cardiology, Mt. Sinai Medical Center, Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ConanTrial
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-08

CONDITIONS: Contrast Induced Nephropathy
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Nitroglycerin (Active Comparator): IV Nitroglycerin with IV Fluids
  Interventions: Drug: Intravenous Nitroglycerin; Drug: IV Fluids
- Placebo (Placebo Comparator): IV Fluids
  Interventions: Drug: IV Fluids

INTERVENTIONS:
Drug: Intravenous Nitroglycerin
  Arms: Intravenous Nitroglycerin
Drug: IV Fluids

SUMMARY:
Contrast-induced nephropathy (CIN) is a complication of percutaneous coronary angiography that occurs in about 10 to 20% of patients exposed to contrast media. Iodinated contrast is used during coronary angiography to see the coronary arteries. It has been shown that exposure to this agent may cause kidney injury. CIN usually goes away on its own but in some high risk patients it progresses into renal failure.

This research study offers a new possible option to prevent CIN. We propose that if intravenous nitroglycerin is given before the procedure it may lower the chances of developing contrast-induced nephropathy.

DETAILED DESCRIPTION:
The Contrast Nephropathy and Nitrates trial (CoNaN) is a single center, randomized, 1 x 1 factorial clinical trial designed to test the effects of intravenous nitroglycerin infusion in renal function given prior to PCI.

Specific aims for this trial include:

* To determine whether the intravenous nitrates have any effect on the glomerular filtration rate (GFR) after the exposure to contrast media.
* To determine if intravenous nitroglycerin will decrease the incidence of contrast induced Nephropathy.

  400 patients with a Mehran score of > 6 and a pre-procedural creatinine measurement will be enrolled. Following baseline assessments, patients will be randomly assigned to receive intravenous infusion nitroglycerine plus intravenous normal saline or normal saline only. Subjects will participate in this study from the time they sign consent (prior to angiographic procedure), until 48-72 hours post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be scheduled for percutaneous coronary angiography.
2. Patients must have a Mehran score more or equal to 6 before the procedure.
3. Patients must have baseline creatinine and hemoblogin drawn before the procedure.
4. Signed informed consent.

Exclusion Criteria:

1. Patients on renal replacement therapy before randomization, will be excluded.
2. Being exposed to any types of nitrates 48 hours prior to randomization,
3. History of allergic reaction to any of the components of intravenous nitroglycerin.
4. Exposure to contrast media 4 days prior randomization.
5. Planned revascularization in the next 24 to 48 hours of the first PCI procedure.
6. The patient is hypotensive (<90/60mmHg) at the time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gervasio Lamas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Nitroglycerin: Intravenous Nitroglycerin with IV Fluids
Period: Overall Study
Arm/Group | Intravenous Nitroglycerin | Placebo
Started | 68 | 54
Completed | 68 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 122 patients consented for participation, met all inclusion/exclusion criteria and were analyzed in the intention-to-treat protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Nitroglycerin | Placebo | Total
Number analyzed (Participants) | 68 | 54 | 122
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 77 [69.5 to 82] | 76 [68 to 85] | 76 [69 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 52 | 38 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 26 | 21 | 47
  Race/Ethnicity: Black | 5 | 3 | 8
  Race/Ethnicity: Asian | 2 | 2 | 4
  Race/Ethnicity: Hispanic | 34 | 27 | 61
  Race/Ethnicity: Unknown/not reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68 | 54 | 122
eGFR (Baseline) [Median (Inter-Quartile Range); unit: mL/min] — estimated Glomerular Filtration Rate
  mL/min | 58.3 [43.7 to 78.5] | 59.1 [48.5 to 77.6] | 58.6 [46.7 to 77.9]

OUTCOME MEASURES:

1. Primary Outcome: Change in GFR
Description: The primary endpoint for this trial will be to determine the change in glomerular filtration rate after exposure to contrast media. We will compare the change in GFR before and after PCI of the group that received intravenous nitroglycerin with the change in GFR before and after PCI of the group that did not receive intravenous nitroglycerin.
Time Frame: Baseline and 48 to 72 hours post-PCI
Measure: Median (Inter-Quartile Range); unit: mL/min
Groups:
- Intravenous Nitroglycerin: IV Nitroglycerin with IV Fluids
  Intravenous Nitroglycerin
  IV Fluids
Arm/Group | Intravenous Nitroglycerin | Placebo
Number analyzed (Participants) | 68 | 54
mL/min | 1.8 [-5.9 to 6.9] | -4.1 [-9.3 to 3]

ADVERSE EVENTS:
Time Frame: 4 years
Description: The collection of adverse events does not differ from the clinicaltrials.gov definitions.
Arm/Group | Intravenous Nitroglycerin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/54
Other Adverse Events (participants affected / at risk) | 4/68 | 2/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Nitroglycerin (N=68) | Placebo (N=54)
Hypotension (Cardiac disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT01999517/Prot_SAP_000.pdf